CLINICAL TRIAL: NCT05355142
Title: Brain Network Mechanism of Pain Empathy and Anhedonia in Patients With Depression by Group Problem Management Plus Intervention
Brief Title: An Intervention Study of Anhedonia and Pain Empathy in Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Fengqiong Yu, Associate Professor, Anhui Medical University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y&H
Record Dates: First submitted 2022-04-18; First posted 2022-05-02 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Treatment Resistant Depression; Problem Management Plus; Event-Related Potentials
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PM+ (Experimental): Intervention once a week for a total of 5 weeks
  Interventions: Behavioral: PM+
- control group (No Intervention): Just daily observation

INTERVENTIONS:
Behavioral: PM+ — 1 Brief introduction to PM+ & NDA (5 min) Assessment-based review with PSYCHOLOPS (psychopomps psychology ) assessment (10 min) What is PM+ (20 minutes) Understanding Adversity (30 minutes) Stress Management (20 minutes) Closing the meeting (5 minutes)
  2 General Review (5 min) Issue management (70 minutes) Stress management (10 minutes) Closing the meeting (5 minutes)
  3 General Review (5 minutes) Problem Management (35 minutes) Take action and be consistent (35 minutes) Stress management (10 minutes) Closing the meeting (5 minutes)
  4 General Review (5 minutes) Issue Management (20 minutes) Take action and be persistent (20 minutes) Strengthening Social Support (30 minutes) Stress management (10 minutes) Closing the meeting (5 minutes)
  5 General Review (20 minutes) Staying Healthy (30 minutes) Imagining how to help someone (20 minutes) Looking ahead (15 minutes) Closing the de-briefing (5 minutes)
  Arms: Group PM+

SUMMARY:
Brain Network Mechanism of Pain Empathy and Anhedonia in Patients With Depression by Group Problem Management Plus Intervention.

DETAILED DESCRIPTION:
It is expected to collect 66 college students.

1. Depressed college students；Healthy control:

   Inclusion criteria: 1) college students; 2) PHQ-9 > 4 points; 2) After informing the content of the study, agree to join the study, sign the informed consent form and accept relevant examination; 3) No major physical diseases in the past; Exclusion criteria: 1) lack of basic data; 2) Those who are currently diagnosed with depression and receiving psychotherapy; 3) Those who are unwilling to accept the inspection and quit halfway; 4) History of brain trauma, or accompanied by serious physical diseases, such as heart and liver dysfunction;
2. Scale evaluation:

   2.1 background information: gender, age, years of education, marriage and childbirth, place of residence (urban and rural), family economic situation (poor, general and good), family structure (core, single parent, reorganization and separation), self-rated learning pressure (high, general and low), whether he is an only child and whether he is a class cadre, etc.

   2.2 depression assessment: Depression Screening Scale (PHQ-9), 2.3 symptom evaluation of loss of pleasure: time experience pleasure scale (TEPS); Loss of social pleasure (RSAs) 2.4 UCLA Loneliness Scale; TAS Alexithymia Scale; Chinese version of interpersonal response index scale (IRI)
3. Experimental paradigm was measured before and after psychological intervention 3.1 Intensive delay First, the subjects were presented with a signal indicating that the cue was 400ms. After cue, the fixation point was 2250-2750 MS, and then the target stimulus square appeared. The presentation time was 160 ms to 260 Ms. The subjects are required to respond to the target stimulation key at the fastest speed. The time of random presentation of fixation is 1450ms. The feedback signal is given according to the results of the subjects' key response, and the presentation time is 1650ms. Finally, the fixation point was presented for 1200-1500ms; The whole paradigm includes two types of reward tasks; One is monetary reward and the other is social reward. Each task consists of 88 trials, resulting in a total of 176 trials.

   3.2 Experimental paradigm of pain empathy In the experiment, the screen first presents a 400ms "+" fixation point, then presents a 400ms empty screen, and then presents a 1000ms picture stimulus. After the stimulus is presented, the empty screen is 1500 ~ 1700ms. The experiment consists of two tasks: ① pain judgment task, which requires subjects to judge whether the body owner in the picture will feel pain ② Left right judgment task: the task requires the subjects to distinguish the left and right limbs in the picture. The subjects also need to watch the picture carefully and make a judgment as quickly and accurately as possible。
4. PM + (problem management plus) intervention is a psychological intervention of 1.5 hours each time for five weeks. Four strategies are mainly taught so that students can use them in daily life. PM + includes four core strategies: (1) decompression (breathing relaxation, mindfulness, etc.); (2) Problem management (coping strategies for practical problems); (3) Act by words, persevere, and emphasize behavior activation (mainly for the strategy of withdrawal of depressive behavior); (4) Strengthen interpersonal relationships (emphasis on strengthening interpersonal connections).

ELIGIBILITY:
Inclusion Criteria:

1. College students;
2. PHQ-9 > 4 points;
3. After informing the content of the study, agree to join the study, sign the informed consent form and accept relevant examination;
4. No major physical diseases in the past;

Exclusion Criteria:

1. Lack of basic data;
2. Those who are currently diagnosed with depression and receiving psychotherapy;
3. Those who are unwilling to accept the inspection and quit halfway;
4. History of brain trauma, or accompanied by serious physical diseases, such as heart and liver dysfunction;

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Patient Health Questionnaire | baseline;5 weeks post-treatment
  The four-level scoring of the PHQ-9 Depression Screening Scale, consisting of nine items with a total score of 0-27, where 0-4 is no depression, 5-9 may have mild depression, 10-14 may have moderate depression, 15-19 may have moderate to severe depression, and 20-27 may have severe depression, has proven validity for application in Chinese adult and college student populations with an internal consistency coefficient of 0.854 and a retest reliability of 0.873.
Change from baseline in Temporal Experience of Pleasure Scale | baseline;5 weeks post-treatment
  The Temporal Experience Pleasure Scale consists of anticipatory (TEPS-anti) and consummatory anhedonia subscales (TEPS-con) with lower scores indicating stronger anhedonia propensity. The Chinese version has demonstrated high internal consistence (Cronbach's alpha = 0.84) .
Change from baseline in Toronto Alexithymia Scale | baseline;5 weeks post-treatment
  The TAS developed by Taylor et al. in 1994 was used, with 20 items on a 5-point scale ranging from "totally disagree" to "totally agree". The scale contains three factors, namely, Disorders of Affective Identification (DIF), Disorders of Descriptive Affect (DDF), and Extraverted Thinking, and the TAS was tested for high reliability and validity.

SECONDARY OUTCOMES:
The change from baseline in behavioral results of Incentive Delay task | baseline; 5 weeks post-treatment change from baseline after the treatment
  The amplitudes of brain potentials of assessed by eventrelated brain potentials methods change from baseline after the treatment.
The change from baseline in event-related brain potentials during Pain empathy task | baseline; 5 weeks post-treatment change from baseline after the treatment
  The amplitudes of brain potentials of assessed by eventrelated brain potentials methods change from baseline after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Kai, MD, Study Chair — Anhui Medical University; Fengqiong Yu, MD, Study Director — Anhui Medical University; Kongliang He, MD, Study Director — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China